CLINICAL TRIAL: NCT01308112
Title: A Randomised Trial to Assess the Safety and Efficacy or Iron Supplementation in Kenyan Pregnant Women
Brief Title: Prenatal Iron and Malaria Study
Acronym: PIMAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Nairobi (Other); Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSHTM-5664
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Malaria
Keywords: Iron; Plasmodium; Malaria; Pregnancy; Kenya
MeSH Terms: conditions — Malaria | interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supplemental iron (Experimental)
  Interventions: Dietary Supplement: iron
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: iron

INTERVENTIONS:
Dietary Supplement: iron — Daily supplementation with iron (60 mg) as ferrous sulphate

SUMMARY:
The purpose of this study is to compare the presence of Plasmodium infection in parturient women who antenatally received a combination of iron-fortified foods with iron supplements versus iron-fortified foods only.

DETAILED DESCRIPTION:
As per recommendations by the World Health Organization (WHO), iron supplementation in children should be restricted in malaria-endemic areas because of concerns that it can lead to an increased burden of malaria. Universal iron supplementation continues to be recommended, however, for women during pregnancy and 3 months postpartum. Observational studies have shown that iron deficiency in parturient women is associated with a marked reduction in the prevalence and density of malarial parasites in the placenta. Plasmodium infections in pregnant women have devastating effects on the foetus and neonate, causing low birth weight, intrauterine growth retardation, preterm delivery, spontaneous abortion, stillbirth and neonatal mortality. Based on our previous work, the Kenyan government is currently drafting legislation for mandatory iron fortification of industrially milled flour. Implementation of the new fortification policy means that pregnant women will receive iron through a combination of fortified foods and supplementation. The investigators are concerned about the safety of the high iron intake resulting from such a policy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 15-45 years resident in the predefined study area
* Pregnant, with gestational age <23 weeks

Exclusion Criteria:

* Failure to provide a blood sample
* Initial haemoglobin concentration <90 g/L
* Reported medical history suggestive of sickle cell anaemia, epilepsy, diabetes
* Obstetric history suggestive of eclampsia or pre-eclampsia
* Obvious mental retardation or metabolic disorder;
* No written consent
* Carrying multiples
* Woman planning to leave the homestead or to be absent for prolonged periods in the course of the pregnancy or within a 1-month period thereafter
* Woman planning to deliver outside the research clinic.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 470 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Maternal Plasmodium infection | Parturition
  Assessed by LDH- and HRP2-based dipstick test and PCR

SECONDARY OUTCOMES:
Serum non-transferrin bound iron concentration | 3 h after ingestion of first supplement with either iron or placebo
Neonatal iron stores | At 1 month of age
  Assessed by plasma ferritin concentration, restricted to infants without inflammation
Maternal iron status | At 1 month after delivery
  To be assessed by haemoglobin concentrations, prevalence of iron deficiency anaemia (plasma ferritin concentration <12 µg/L) and iron stores (ratio of ferritin:transferrin receptor concentrations); indicators based on ferritin and/or transferrin receptor will be restricted to those without inflammation.
Maternal intestinal pathogens | At 1 month after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Hans Verhoef, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- University of Nairobi, Nairobi, Kenya

REFERENCES:
- [Derived] Mwangi MN, Roth JM, Smit MR, Trijsburg L, Mwangi AM, Demir AY, Wielders JP, Mens PF, Verweij JJ, Cox SE, Prentice AM, Brouwer ID, Savelkoul HF, Andang'o PE, Verhoef H. Effect of Daily Antenatal Iron Supplementation on Plasmodium Infection in Kenyan Women: A Randomized Clinical Trial. JAMA. 2015 Sep 8;314(10):1009-20. doi: 10.1001/jama.2015.9496. PMID 26348751
- [Derived] Mwangi MN, Maskey S, Andang o PE, Shinali NK, Roth JM, Trijsburg L, Mwangi AM, Zuilhof H, van Lagen B, Savelkoul HF, Demir AY, Verhoef H. Diagnostic utility of zinc protoporphyrin to detect iron deficiency in Kenyan pregnant women. BMC Med. 2014 Nov 26;12:229. doi: 10.1186/s12916-014-0229-8. PMID 25428714